CLINICAL TRIAL: NCT00528476
Title: Role of Clinical and Urodynamic Risk Factors for Recurrent Urinary Tract Infection in 5-18 Years Old Children
Brief Title: Risk Factors for Recurrent Urinary Tract Infection in Children
Status: Completed | Type: Observational
Sponsor: Kaunas University of Medicine (Other)
Other Study IDs: BE-2-68
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Last update posted 2007-09-12 (Estimated); Status verified 2007-09

CONDITIONS: Urinary Tract Infection; Pyelonephritis; Cystitis
Keywords: pyelonephritis; cystitis; risk factor; children; urodynamics
MeSH Terms: conditions — Urinary Tract Infections; Pyelonephritis; Cystitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients, who were treated because of recurrent (2 or more urinary tract infections per year) pyelonephritis or cystitis.
- 2: Patients with nonrecurrent urinary tract infections (patients who had no history of more than one urinary tract infections in last year).

SUMMARY:
The purpose of this study is to determine clinical and urodynamic risk factors for recurrent urinary tract infection in 5-18 years old children.

DETAILED DESCRIPTION:
It is known, that in the group of young children the most common reason of recurrent UTI is anatomic abnormalities, such as vesicoureteral reflux, hydronephrosis. However, not all recurrent UTI can be explained by anatomic abnormalities. The vast majority of school age children with recurrent UTI have anatomically normal urinary tract. Recent studies discuss about the role of behavioral and functional abnormalities (inadequate fluid intake, stool retention, infrequent voiding, etc.) that can predispose recurrent urinary tract infections. Influence of some these abnormalities for recurrent UTI is controversial. Family history, behavioral and functional abnormalities which predispose to urinary tract infections in children with normal urinary tract are neglected in most protocols of urinary tract infection.

Children in this study receive a careful evaluation including complete history, voiding-drinking diary, bowel questionnaire, physical investigation, sonography, voiding cystourethrogram.

Follow up time - 1 year. Urinalysis once a month and during each episode of fever.

ELIGIBILITY:
Inclusion Criteria:

* 5-18 years old children, who were treated because of cystitis and pyelonephritis in Kaunas Medical University Hospital

Exclusion Criteria:

* urinary tract malformations
* neurogenic bladder dysfunction
* patients, who received immunosuppressive drugs
* pregnant girls
* children with non bacterial urinary tract infection

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 161 (Actual)
Dates: Start 2004-11; Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarunas Rudaitis, MD, Principal Investigator — Clinic of Children's Diseases, Kaunas University of Medicine; Birute Pundziene, MD, PhD, Study Chair — Clinic of Children's Diseases, Kaunas University of Medicine
Locations (1):
- Kaunas University of Medicine, Kaunas, Lithuania